CLINICAL TRIAL: NCT07304960
Title: Comparative Study Between Multiple Sclerosis Versus Neuromyelitis Optica Spectrum Disorder Patients in Assiut Hospitals Clinical and Laboratory Study
Brief Title: Multiple Sclerosis Versus Neuromyelitis Optica Spectrum Disorder
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hussein Abd Elrahim Hussein Mohamed, Resident doctor, Assiut University
Other Study IDs: MS VS NMO-2026
Record Dates: First submitted 2025-11-27; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: MS (Multiple Sclerosis); NMO Spectrum Disorder (NMOSD)
MeSH Terms: conditions — Multiple Sclerosis; Neuromyelitis Optica

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this work is to do a detailed comparison between multiple sclerosis and Neuromyelitis Optica Spectrum Disorder due to delicate similarities between both diseases and wide rang of management and follow up of the patients

ELIGIBILITY:
Inclusion Criteria:1- Both sex 2- Aged between 18 and 50 years. All included patients were in a clinically stable phase and had not experienced a relapse within at least three months before blood sampling. 3- All patients diagnosed as MS patients either naive or on disease modifying therapies according to The new diagnostic criteria MacDonalds 2024 4- DMT-naïve NMOSD patients: Diagnosed with MS based on the 2017 McDonald Criteria (Thompson et al., 2018)

5- An informed consent will be obtained from all the patients; the study will be approved by ethical committee in faculty of Medicine Assiut University

-

1_ Presence of other disorder that mimic MS or NMOSD 3_ Patients failed to commit to the follow up visits and regular MRI scans 4_ Patients refused to sign the written informed consent

Exclusion Criteria:

* 1_ Presence of other disorder that mimic MS or NMOSD 3_ Patients failed to commit to the follow up visits and regular MRI scans 4_ Patients refused to sign the written informed consent

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: Patients attending toassuit hospitals
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2030-12-22 (Estimated); Study Completion 2030-12-22 (Estimated)

PRIMARY OUTCOMES:
serum Glial Fibrillary Acidic Protein levels | Baseline
  Measurement of serum concentrations of Glial Fibrillary Acidic Protein at baseline using a validated immunoassay (e.g., single-molecule array [Simoa] assay). difference in serum Glial Fibrillary Acidic Protein levels between treatment-naïve NMOSD and treatment-naïve MS patientsexpressed in picograms per milliliter (pg/mL).

SECONDARY OUTCOMES:
Correlation between serum biomarkers (sGFAP and sNfL) and lesion burden on MRI. | Baseline
  Correlation (Pearson or Spearman) between biomarker levels and total T2 lesion count at baseline MRI.
Correlation between serum biomarkers (sGFAP and sNfL) and Expanded Disability Status Scale (EDSS). | Baseline
  Correlation analysis (Pearson or Spearman depending on distribution) between baseline serum concentrations of sGFAP/sNfL and baseline EDSS scores.
Association between serum biomarkers and optic nerve involvement (length and presence of LETM). | Baseline
  Correlation between sGFAP/sNfL levels and MRI-measured optic nerve lesion length, including presence of longitudinally extensive transverse myelitis (LETM).
Diagnostic performance of sGFAP and combined sGFAP + sNfL in differentiating NMOSD from MS. | Baseline
  Assessment of diagnostic accuracy using Area Under the Receiver Operating Characteristic Curve (AUC) for:
  1. sGFAP alone
  2. Combined biomarker model (sGFAP + sNfL)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lublin FD, Reingold SC, Cohen JA, Cutter GR, Sorensen PS, Thompson AJ, Wolinsky JS, Balcer LJ, Banwell B, Barkhof F, Bebo B Jr, Calabresi PA, Clanet M, Comi G, Fox RJ, Freedman MS, Goodman AD, Inglese M, Kappos L, Kieseier BC, Lincoln JA, Lubetzki C, Miller AE, Montalban X, O'Connor PW, Petkau J, Pozzilli C, Rudick RA, Sormani MP, Stuve O, Waubant E, Polman CH. Defining the clinical course of multiple sclerosis: the 2013 revisions. Neurology. 2014 Jul 15;83(3):278-86. doi: 10.1212/WNL.0000000000000560. Epub 2014 May 28. PMID 24871874
- [Result] Wingerchuk DM, Banwell B, Bennett JL, Cabre P, Carroll W, Chitnis T, de Seze J, Fujihara K, Greenberg B, Jacob A, Jarius S, Lana-Peixoto M, Levy M, Simon JH, Tenembaum S, Traboulsee AL, Waters P, Wellik KE, Weinshenker BG; International Panel for NMO Diagnosis. International consensus diagnostic criteria for neuromyelitis optica spectrum disorders. Neurology. 2015 Jul 14;85(2):177-89. doi: 10.1212/WNL.0000000000001729. Epub 2015 Jun 19. PMID 26092914
- [Result] Thompson AJ, Banwell BL, Barkhof F, Carroll WM, Coetzee T, Comi G, Correale J, Fazekas F, Filippi M, Freedman MS, Fujihara K, Galetta SL, Hartung HP, Kappos L, Lublin FD, Marrie RA, Miller AE, Miller DH, Montalban X, Mowry EM, Sorensen PS, Tintore M, Traboulsee AL, Trojano M, Uitdehaag BMJ, Vukusic S, Waubant E, Weinshenker BG, Reingold SC, Cohen JA. Diagnosis of multiple sclerosis: 2017 revisions of the McDonald criteria. Lancet Neurol. 2018 Feb;17(2):162-173. doi: 10.1016/S1474-4422(17)30470-2. Epub 2017 Dec 21. PMID 29275977
- [Result] Rae-Grant A, Day GS, Marrie RA, Rabinstein A, Cree BAC, Gronseth GS, Haboubi M, Halper J, Hosey JP, Jones DE, Lisak R, Pelletier D, Potrebic S, Sitcov C, Sommers R, Stachowiak J, Getchius TSD, Merillat SA, Pringsheim T. Practice guideline recommendations summary: Disease-modifying therapies for adults with multiple sclerosis: Report of the Guideline Development, Dissemination, and Implementation Subcommittee of the American Academy of Neurology. Neurology. 2018 Apr 24;90(17):777-788. doi: 10.1212/WNL.0000000000005347. PMID 29686116